CLINICAL TRIAL: NCT06266143
Title: Phase Ib/II Trial of Y101D Combined With Gemcitabine and Albumin Paclitaxel in First-line Treatment of Patients With Advanced Pancreatic Cancer
Brief Title: A Trial of Y101D in Combination With Gemcitabine and Albumin Paclitaxel in Patients With Advanced Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wuhan YZY Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y101D03
Record Dates: First submitted 2024-01-24; First posted 2024-02-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Advanced Pancreatic Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): Y101D combined with Gemcitabine and Nab-Paclitaxel
  Interventions: Drug: Y101D

INTERVENTIONS:
Drug: Y101D — Intravenous infusion of Y101D at day1, combined with Gemcitabine and Nab-Paclitaxel IV infusion at day1, 8, a 21-day cycle. After 6 cycles, Y101D and Gemcitabine infusion is applied as the maintenance treatment.

SUMMARY:
The Phase Ib/II study is an open-label, single-arm, multicenter trial designed to assess the efficacy and safety of Y101D in combination with Gemcitabine and Albumin Paclitaxel as first-line systemic treatment for advanced pancreatic cancer patients. The Phase Ib portion of the study aims to evaluate the safety of escalating doses of Y101D in combination with the standard regimen of Gemcitabine and Albumin Paclitaxel and determine the recommended phase 2 dose (RP2D). The Phase II portion of the study aims to evaluate the effectiveness of this combination treatment in a small population of patients.

DETAILED DESCRIPTION:
A total of 57-81 systemic treatment-naïve patients with advanced pancreatic cancer will be enrolled in the study. Phase Ib will enroll 12-36 patients to assess the safety of Y101D combined with Gemcitabine and Albumin Paclitaxel at doses of 20mg/kg or 30mg/kg. The recommended phase 2 dose (RP2D) for Y101D in combination with the other drugs will be determined based on the safety profile and preliminary efficacy data.

Following determination of the RP2D, Phase II will enroll a total of 40-45 patients to evaluate the effectiveness of the combination treatment using the RP2D of Y101D. The primary endpoint of the Phase II study will be the objective response rate. Secondary endpoints will include progression-free survival (PFS), overall survival (OS), duration of response (DOR) and safety profiles. Pharmacodynamic parameters such as serum tumor biomarkers and TGF-β concentration will also be evaluated.

Overall, the study aims to assess the safety, efficacy, and pharmacodynamics of Y101D in combination with Gemcitabine and Albumin Paclitaxel as a first-line systemic treatment for advanced pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pancreatic cancer (including ductal adenocarcinoma and acinar cell carcinoma) confirmed by histology or cytology; and evidence of unresectable or distant metastasis.
* No prior systemic treatment for advanced/metastatic pancreatic cancer.
* Previous use of anti-tumor Chinese herbal medicine or traditional Chinese medicine preparations, but discontinued use at least 28 days before the first administration of the investigational drug.
* According to RECIST 1.1 criteria, the subject must have at least one measurable target lesion confirmed by CT or MRI examination that has not been locally treated (unless the target lesion has clearly progressed).
* Expected survival time ≥ 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
* According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, any toxicity from previous anti-tumor treatment or surgery must have recovered to grade 0-1 or to the level specified by the inclusion/exclusion criteria. Note: Exclusions include alopecia, pigmentation changes, ≤ grade 2 neuropathy, hypothyroidism due to hormone replacement, or other adverse events confirmed to have become chronic.
* Organ function levels must meet the following requirements:

Hematology: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, lymphocyte count ≥ 0.5 × 109/L, platelets (PLT) ≥ 100 × 109/L, hemoglobin (HGB) ≥ 90g/L (within 14 days before screening without blood transfusion, use of blood products, or correction with granulocyte colony-stimulating factor [G-CSF] or other hematopoietic growth factors).

Liver function: Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal, aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 times the upper limit of normal (if there is liver metastasis, AST and ALT up to 5 times the upper limit of normal are allowed).

Renal function: Serum creatinine (Cr) ≤ 1.5 times the upper limit of normal or creatinine clearance rate ≥ 50 mL/min (Cockcroft-Gault formula).

Coagulation function: International normalized ratio (INR) ≤ 1.5, prothrombin time (PT), and activated partial thromboplastin time (APTT) ≤ 1.5 times the upper limit of normal.

Exclusion Criteria:

* Patients diagnosed with central nervous system (CNS) metastasis confirmed by imaging.
* Patients with diseases associated with a high risk of clinically significant gastrointestinal bleeding (such as tumor invasion of the gastrointestinal tract or bile ducts) or any other condition or history related to severe bleeding.
* Presence of clinically uncontrollable third-space fluid accumulation before the first administration of the investigational drug, such as pleural effusion, ascites, or pericardial effusion that cannot be controlled by drainage or other methods, as determined by the investigator.
* Underwent major surgery within 4 weeks prior to the first administration of the investigational drug (excluding needle biopsies and tooth extractions).
* Use of immunosuppressive drugs within 7 days prior to the first administration of the investigational drug, excluding nasal and inhaled corticosteroids or physiological doses of systemic corticosteroid hormones
* Significant clinical pancreatitis.
* History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Presence of active clinical infection of grade 2 or higher (according to CTCAE v5.0 criteria) at screening, requiring systemic (oral or intravenous) antimicrobial treatment.
* Patients requiring long-term use of steroids or immunosuppressive agents for conditions such as active autoimmune diseases or post-organ transplant maintenance therapy. Exceptions include type 1 diabetes, hypothyroidism that can be controlled by replacement therapy alone, and skin diseases (such as vitiligo, psoriasis, or alopecia) that do not require systemic treatment.
* Severe respiratory system diseases or patients judged by the investigator to be unsuitable for inclusion, or patients with concomitant interstitial pneumonia.
* Average corrected QT interval (QTcF) >450 msec (males) or >470 msec (females) based on three electrocardiogram (ECG) examinations during screening (repeat testing and averaging of three measurements are required only if the first ECG indicates QTcF >450 msec [males] or >470 msec [females]). History of long or short QT syndrome in the family or individual, or significant cardiovascular diseases within 6 months before screening.
* History of non-study malignancy (excluding non-invasive lesions with extremely low risk of recurrence, such as squamous cell carcinoma and basal cell carcinoma of the skin, cervical carcinoma in situ, or breast carcinoma in situ) within 5 years prior to the first administration of the investigational drug.
* Active hepatitis B (positive hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb], peripheral blood HBV DNA titers <500 IU/mL allow inclusion), active hepatitis C, active syphilis, HIV-positive patients.
* Pregnant or lactating women, or individuals with reproductive potential within 6 months after the end of this clinical study, regardless of gender.
* Known history of substance abuse or drug addiction.
* History of clear neurological or psychiatric disorders, as determined by the investigator, that would hinder compliance with treatment or adherence to instructions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | From the time of the first dose (Day 1) until Day 21
  Dose limiting toxicities during the first 21 days after the first administrations of Y101D in each cohort.
RP2D | From the enrollment of first patient through phae 1b study completion, an average of 1 year
  Recommended Phase 2 Dose of Y101D
Objective Response Rate (ORR) | From the time of first dosing (Day 1) until disease progression (up to 6 months)
  Objective Response Rate assessed according to RECIST 1.1 per investigator

SECONDARY OUTCOMES:
Peak Serum Concentration (Cmax) | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months).
  The highest Y101D concentration in serum during one treatment cycle (21 days)
Trough Serum Concentration (Ctrough) | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months).
  The lowest Y101D concentration in serum during one treatment cycle (21 days)
Area under the serum concentration versus time curve (AUC) during one treatment cycle (21 days) | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months).
  The area under the serum concentration versus tiem curve of Y101D during one treatment cycle (21 days)
The TGF-β concentration in serum | From the time of first dosing (Day 1) until disease progression or death or toxicity intolerance (up to 6 months).
  The TGF-β concentreation in serum at 30 minutes before the first treatment dosing of Y101D and the subsequent dosing of Y101D every two cycles (Cycle 3 Day 1, Cycle 5 Day 1, etc.) until the disease progression or death or toxicity intolerance of Y101D.
The CA19-9 concentration in serum | From the time of first dosing (Day 1) until disease progression or death or toxicity intolerance (up to 6 months).
  The CA19-9 concentreation in serum at 30 minutes before the first treatment dosing of Y101D and the subsequent dosing of Y101D every two cycles (Cycle 3 Day 1, Cycle 5 Day 1, etc.) until the disease progression or death or toxicity intolerance of Y101D.
The positive rate of Anti-Drug Antibody (ADA) and Neutralizing antibody (Nab) | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months)
  The potivie rate of Anti-Drug Antibody and neutralizing antibody in serum 30 minutes before the Y101D infusion at Day 1 of Cycle 1, Cycle 2, Cycle 4 and Cycle 7 (a 21-day cycle).
Disease control rate (DCR) | From the time of first dosing (Day 1) until disease progression or toxicity intolerance (up to 6 months).
  Disease control rate assessed according to RECIST 1.1 per investigator
Duration of response (DOR) | From the time of first dosing (Day 1) until one month after the EOT
  The time from the first objective response to disease progression or death
Progression-free survival (PFS) | From the time of first dosing (Day 1) until disease progression or death (up to 12 months).
  The time from the first objective response to disease progression or death (Up to 12 months)
Overall survival (OS) | From the time of first dosing (Day 1) until death (up to 2 years).
  The time from the first objective response to death (Up to 2 yrs)

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No